CLINICAL TRIAL: NCT01244360
Title: The Effects of Resveratrol Supplementation on Measurements of Health and Human Performance
Acronym: MUresv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marywood University (Other)
Responsible Party: JAmes Smoliga, Ph.D., Marywood University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU Smoliga Resveratrol; 2RESMU194218 (Other: Marywood University)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Inflammation
Keywords: resveratrol; insulin; inflammation; cognition; metabolism
MeSH Terms: conditions — Inflammation; Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Subject will take placebo for daily for 4 weeks, with optional additional 4 week treatment period.
  Interventions: Other: Placebo Comparator: Sugar Pill
- Dietary Supplement: resveratrol (Active Comparator): Subject will take resveratrol supplement for 4 weeks, with optional additional 4 week treatment period.
  Interventions: Dietary Supplement: resveratrol

INTERVENTIONS:
Dietary Supplement: resveratrol — Subject will take resveratrol supplement for 4 weeks, with optional additional 4 week treatment period.
  Arms: Dietary Supplement: resveratrol
Other: Placebo Comparator: Sugar Pill — Subject will take placebo for daily for 4 weeks, with optional additional 4 week treatment period.
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to examine the effects of resveratrol on health and human performance. The study will evaluate cognitive function and several indicators of physical health before and after taking a resveratrol supplement or a placebo for three weeks.

DETAILED DESCRIPTION:
Measurements

* blood laboratory parameters
* cognitive assessment changes
* body composition changes
* vascular endothelial response

ELIGIBILITY:
Inclusion Criteria:

* men and women between 45 and 75 years of age
* Normal heart rate and Blood pressure
* Ability to use personal computer interface
* Successful completion of physical activity readiness questionnaire

Exclusion Criteria:

* Cardiovascular disease, uncontrolled hypertension, lung disease
* inability to tolerate exercise
* have taken grape related supplement in past 12 months
* current use of drugs or dietary supplements to enhance exercise performance
* allergy to wine, grape juice or grape seed supplements

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Vascular function | 4 weeks, with option of additional 4 week treatment period
  vascular response to stress will be measured using flow mediated dilation and ultrasound.

SECONDARY OUTCOMES:
Body fat percentage | 4 weeks, with optional additional 4 week treatment period
  Body fat percentage will be measured using a DEXA scan.
inflammation biomarkers | 4 weeks, with optional additional 4 week treatment period
  Fasting blood draw
cognitive function | 4 weeks, with optional additional 4 week treatment period
  cognitive function will be assessed using a validated computer based assessment tool

CONTACTS AND LOCATIONS:
Overall Officials: James Smoliga, Ph.D., Principal Investigator — Marywood University
Locations (1):
- Marywood University, Scranton, Pennsylvania, United States